CLINICAL TRIAL: NCT03465423
Title: Comparison of Propofol Requirement Between Patients With Pituitary Somatotroph Tumor and With Nonfunctioning Pituitary Tumor in Transsphenoidal Pituitary Surgery Under Total Intravenous Anesthesia
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-1241
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pituitary Tumor
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with nonfunctioning pituitary tumor: patients with nonfunctioning pituitary tumor undergoing transsphenoidal pituitary surgery under total intravenous anesthesia
  Interventions: Procedure: Not applicable (measuring subject's effect site concentration of propofol during the induction of general anesthesia)
- patients with pituitary somatotroph tumor: patients with pituitary somatotroph tumor undergoing transsphenoidal pituitary surgery under total intravenous anesthesia
  Interventions: Procedure: Not applicable (measuring subject's effect site concentration of propofol during the induction of general anesthesia)

INTERVENTIONS:
Procedure: Not applicable (measuring subject's effect site concentration of propofol during the induction of general anesthesia) — The patients of two cohort group will undergo general anesthesia in the same way and therefore there is no intervention in this study.

SUMMARY:
Investigators hypothesized that propofol dose for pituitary somatotroph patients might differ from nonfunctioning pituitary tumor, and investigators will evaluate a target controlled infusion (TCI) effect site concentration (Ce) of propofol for BIS score of 40 and LOC (loss of consciousness) in pituitary somatotroph patients in comparison with non functioning pituitary tumor patients.

On arrival in the operating room, standard monitoring devices, including electrocardiogram, pulse oximetry, noninvasive blood pressure cuff, and bispectral index (BIS) will be applied to the patients. Propofol with the modified Marsh pharmacokinetic parameters using a keo of 1.2/min will be administered through TCI pump (OrchestraBase Primea, Fresenius Vial, France). The initial target Ce of propofol will be chosen as 3.0 mg/mL (0.5 mg/mL of incremental size) based on an earlier study.

The sedation of patients will be assessed with BIS score and the modified observer's assessment of awareness and sedation (OAA/S). LOC was defined as an OAA/S lower than 2 (loss of response to spoken command to eye opening and loss of response to mild prodding or shaking). The primary end point of this study is the Ce of propofol when the BIS score is 40. The secondary end point of this study is the Ce of propofol at LOC.

ELIGIBILITY:
Inclusion Criteria:

* patients with pituitary somatotroph tumor and with nonfunctioning pituitary tumor in transsphenoidal pituitary surgery
* American society of anesthesiologists classification 1 or 2

Exclusion Criteria:

* left ventricle ejection fraction < 55% 3RD degree AV block, 2nd degree AV block with P:QRS > 3:1
* serum Creatinine > 1.0mg/dl
* myocardial infarction or cerebral stroke in 1 yrs
* fever > 38C
* dementia, cognitive disorder, confused mental status
* pregnant patients
* allergic to propofol
* illiteracy or foreigners

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Investigators hypothesized that propofol dose for pituitary somatotroph patients might differ from nonfunctioning pituitary tumor, and we will evaluate a target controlled infusion (TCI) effect site concentration (Ce) of propofol for BIS score of 40 and LOC (loss of consciousness) in pituitary somatotroph patients in comparison with non functioning pituitary tumor patients.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
effect site concentration of propofol | 5 minutes after subject's anesthesia induction
  Investigators will assess the propofol requirement in pituitary tumor patients during the induction of general anesthesia when subject's BIS (Bispectral Index Score) is 40

SECONDARY OUTCOMES:
effect site concentration of propofol | 2 minutes after subject's anesthesia induction
  Investigators will assess the propofol requirement in pituitary tumor patients during the induction of general anesthesia when the pituitary tumor patients lose their consciousness.

CONTACTS AND LOCATIONS:
Locations (1):
- Associate Professor Department of Anesthesiology and Pain Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No